CLINICAL TRIAL: NCT04788836
Title: How Altered Gut-Brain-Axis Influences Food Choices. (BrainFood) Part 2: Digital Receipts
Brief Title: How Altered Gut-Brain-Axis Influences Food Choices: Part 2 (BrainFood)
Acronym: BrainFood
Status: Active, not recruiting | Type: Observational
Sponsor: Lia Bally (Other)
Collaborators: ETH Zurich (Other)
Responsible Party: Sponsor-Investigator, Lia Bally, Professor, Insel Gruppe AG, University Hospital Bern
Organization: Insel Gruppe AG, University Hospital Bern (Other)
Other Study IDs: BrainFood Part 2
Record Dates: First submitted 2021-01-18; First posted 2021-03-09 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Food Preferences; Obesity
Keywords: Bariatric surgery; Food preferences; Food behaviour; Digital receipts; Grocery Shopping; Obesity treatment; GLP-1 receptor agonist
MeSH Terms: conditions — Food Preferences; Obesity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Obesity treatment Group: 60 (minimum) to 150 (maximum) overweight/obese adults referred for or who started obesity (surgical or non-surgical) treatment within 6 months
  Interventions: Other: Questionnaire (Survey and Food Frequency Questionnaire (FFQ)); Other: Collection of digital receipts from grocery shopping
- Control Group: Comparison of food purchase behaviour with control subjects will be performed using an already existing cohort from a previous study. This does not required recruiting control subjects.

INTERVENTIONS:
Other: Questionnaire (Survey and Food Frequency Questionnaire (FFQ)) — Each participant will be asked to fill a web-based questionnaire that captures sociodemographic, lifestyle, physical and mental health information (Survey) and dietary intake patterns (FFQ). This will be done pre-treatment (only for those included pre-treatment), 6 months after the start of obesity treatment, 1 year after the start of the treatment and then yearly until 5 year after the start of the treatment.
  Groups: Obesity treatment Group
Other: Collection of digital receipts from grocery shopping — Participants will create their BitsaboutMe-account (GDPR-compliant data sharing platform from Bern, Switzerland) with the help of study team members. Data from digital receipts will be obtained from Migros Cumulus and Coop Supercard via their BitsaboutMe-account. The data collection allow retrospective digital receipts collection for up to 2 years and automatically continuous collection during study duration.
  GDPR: General Data Protection Regulation
  Groups: Obesity treatment Group

SUMMARY:
Obesity is currently one of the most substantial health burdens. Due to the production of marked and sustained weight loss, bariatric surgery is an increasingly used therapeutic modality to combat obesity and its comorbidities. Surgical rearrangement of the gastrointestinal tract remarkably alters metabolism and hormones acting on neurological and hypothalamic signalling, involved in food decision-making and eating behaviour. In this context, many patients who underwent bariatric surgery self-report changes in appetite, satiety and food preferences. Furthermore, new gut hormone-based (e.g. GLP-1 receptor agonist or GLP-1-RA) pharmacotherapies which mimic the effect of bariatric surgery show impressive efficacy on weight reduction by modulation of food behaviour. However, the mechanisms of such functional changes, and how they relate to food decision-making and food purchase behaviour remain unknown.

In Part 2 of the BrainFood-project, the investigators propose a novel approach using digital receipts from loyalty card to unravel the effect of obesity treatments (surgical and non-surgical) on eating and food purchase behaviour in daily life.

DETAILED DESCRIPTION:
The overall aim of this project is to elucidate the changes in food behaviour among obese adults undergoing obesity treatments.

The main objective is to observe the effect of obesity treatments on food purchase behaviour using digital receipts from grocery shopping. The investigators hypothesize that bariatric surgery leads to changes in food purchase behaviour in obese adults.

The further objective is to compare food purchase behaviour between obese adults against values of an existing reference population, and to assess whether these differences tend to be reduced after the start of the treatment among obese participants.

ELIGIBILITY:
Inclusion Criteria:

* Female and male subjects aged 18 years or older
* Proficient in German (including written)
* BMI≥30kg/m2 or BMI≥28kg/m2 with adiposity-related comorbidities (prediabetes, type 2 diabetes mellitus, hypertension, dyslipidemia)
* Referred for obesity treatment or who started obesity treatment within 6 months (surgical or non-surgical)
* Primary grocery shopping at the Swiss biggest grocery retailers (Coop, Migros), and regularly using a loyalty card (Cumulus and/or Supercard)

Exclusion Criteria:

* Incapacity to give informed consent
* Primary shopping in other food retailers (e.g. Aldi, Lidl, outside of Switzerland, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A minimum of 60 (up to a maximum of 150) overweight/obese adults planned for or who started surgical or non-surgical obesity treatment within the past 6 months will be recruited for this study. Participants will be recruited by referral from our outpatient endocrine clinic and collaborating Centres of Excellence for Metabolic Surgery.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes in food purchase behaviour on the basis of the Healthy Trolley Index (HETI) | Pre-treatment until 5 years after start of obesity treatment
  Changes in food purchase behaviour pre-treatment will be compared to post-treatment on the basis of the HETI, an objective and validated, nutrient-based, healthy shopping scoring system.
Changes in food purchase behaviour on the basis of the Grocery Purchase Quality Index (GPQI) | Pre-treatment until 5 years after start of obesity treatment
  Changes in food purchase behaviour pre-treatment will be compared to post-treatment on the basis of the GPQI, an objective and validated, nutrient-based, healthy shopping scoring system.
Changes in food purchase behaviour on the basis of food groups | Pre-treatment until 5 years after start of obesity treatment
  Changes in food purchase behaviour pre-treatment will be compared to post-treatment on the basis of food groups like vegetables, wholegrain, fruits, sweets and meats.
Changes in food purchase behaviour on the basis of nutrition facts | Pre-treatment until 5 years after start of obesity treatment
  Changes in food purchase behaviour pre-treatment will be compared to post-treatment on the basis of nutrition facts like energy (kcal), carbohydrates, sugars, added sugars, protein, fat, saturated fat, dietary fibre and salt.
Changes in food purchase behaviour on the basis of the Nutri-Score | Pre-treatment until 5 years after start of obesity treatment
  Changes in food purchase behaviour pre-treatment will be compared to post-treatment on the basis of the Nutri-Score, representing the nutritional quality of products. The Nutri-Score is based on a discrete continuous scale from -15 (most healthy) to 40 (least healthy). The score is then transcribed into five colour categories (A-E, ranging from bright green (most healthy) to red (least healthy)).
Food purchase behaviour on the basis of the Healthy Trolley Index (HETI) | Pre-treatment until 5 years after start of obesity treatment
  HETI will be compared between obesity treatment group and control group
Food purchase behaviour on the basis of the Grocery Purchase Quality Index (GPQI) | Pre-treatment until 5 years after start of obesity treatment
  GPQI will be compared between obesity treatment group and control group
Food purchase behaviour on the basis of food groups | Pre-treatment until 5 years after start of obesity treatment
  Food groups will be compared between obesity treatment group and control group
Food purchase behaviour on the basis of nutrition facts | Pre-treatment until 5 years after start of obesity treatment
  Nutrition facts will be compared between obesity treatment group and control group
Food purchase behaviour on the basis of the Nutri-Score | Pre-treatment until 5 years after start of obesity treatment
  Nutri-Score will be compared between obesity treatment group and control group

OTHER OUTCOMES:
Correlation between food purchase patterns (i.e. HETI, GPQI, food groups, nutrition facts, Nutri-Score) and self-perceived quality of life | Pre-treatment until 5 years after start of obesity treatment
  Quality of life will be assessed using on a scale from 1 (very bad) to 5 (very good)
Changes in energy intake | Pre-treatment until 5 years after start of obesity treatment
  Energy intake in kilocalories (kcal)/day based on Food Frequency Questionnaire
Changes in daily carbohydrate intake | Pre-treatment until 5 years after start of obesity treatment
  Dietary intake in gram/day based on Food Frequency Questionnaire
Changes in daily sugar intake | Pre-treatment until 5 years after start of obesity treatment
  Dietary intake in gram/day based on Food Frequency Questionnaire
Changes in daily fibre intake | Pre-treatment until 5 years after start of obesity treatment
  Dietary intake in gram/day based on Food Frequency Questionnaire
Changes in daily protein intake | Pre-treatment until 5 years after start of obesity treatment
  Dietary intake in gram/day based on Food Frequency Questionnaire
Changes in daily fat intake | Pre-treatment until 5 years after start of obesity treatment
  Dietary intake in gram/day based on Food Frequency Questionnaire
Changes in daily saturated fat intake | Pre-treatment until 5 years after start of obesity treatment
  Dietary intake in gram/day based on Food Frequency Questionnaire
Changes in daily sodium intake | Pre-treatment until 5 years after start of obesity treatment
  Dietary intake in milligram/day based on Food Frequency Questionnaire
Changes in daily vegetable intake | Pre-treatment until 5 years after start of obesity treatment
  Dietary intake in gram/day based on Food Frequency Questionnaire
Changes in daily wholegrain intake | Pre-treatment until 5 years after start of obesity treatment
  Dietary intake in gram/day based on Food Frequency Questionnaire
Changes in daily fruit intake | Pre-treatment until 5 years after start of obesity treatment
  Dietary intake in gram/day based on Food Frequency Questionnaire
Changes in daily dessert intake | Pre-treatment until 5 years after start of obesity treatment
  Dietary intake in gram/day based on Food Frequency Questionnaire
Changes in daily meat intake | Pre-treatment until 5 years after start of obesity treatment
  Dietary intake in gram/day based on Food Frequency Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lia Bally, MD, PhD, Principal Investigator — University Hospital Bern & University of Bern
Locations (1):
- Department of Diabetes, Endocrinology, Clinical Nutrition and Metabolism, Inselspital, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided